CLINICAL TRIAL: NCT04358536
Title: Classification of COVID-19 Infection in Posteroanterior Chest X-rays With Common Deep Learning Architectures
Brief Title: Classification of COVID-19 Infection in Posteroanterior Chest X-rays
Status: Completed | Type: Observational
Sponsor: Dascena (Industry)
Responsible Party: Sponsor
Other Study IDs: 04202002
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: machine learning; X-ray; classification; COVID-19; posteroanterior; convolutional neural network architectures
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Patients: Single posteroanterior (or "front-on") X-rays collected from COVID-19 patients
  Interventions: Device: CovX
- Non COVID-19 Patients: Single posteroanterior (or "front-on") X-rays collected from subsets of non COVID-19 patients
  Interventions: Device: CovX

INTERVENTIONS:
Device: CovX — Convolutional neural network for classification of COVID-19 from chest X-rays

SUMMARY:
The objective of this study is to assess three configurations of two convolutional deep neural network architectures for the classification of COVID-19 PCX images.

DETAILED DESCRIPTION:
The December 2019 outbreak of COVID-19 has now evolved into a public health emergency of global concern. Given the rapid spread of infection, the rapid depletion of hospital resources due to high influxes of patients, and the current absence of specific therapeutic drugs and vaccines for treatment of COVID-19 infection, it is essential to detect onset of the disease at its early stages. Radiological examinations, the most common of which are posteroanterior chest X-ray (PCX) images, play an important role in the diagnosis of COVID-19. The objective of this study is to assess three configurations of two convolutional deep neural network architectures for the classification of COVID-19 PCX images. The primary experimental dataset consisted of 115 COVID-19 positive and 115 COVID-19 negative PCX images, the latter comprising roughly equally many pneumonia, emphysema, fibrosis, and healthy images (230 total images). Two common convolutional neural network architectures were used, VGG16 and DenseNet121, the former initially configured with off-the-shelf (OTS) parameters and the latter with either OTS or exclusively X-ray trained (XRT) parameters. The OTS parameters were derived from training on the ImageNet dataset, while the XRT parameters were obtained from training on the NIH chest X-ray dataset, ChestX-ray14. A final, densely connected layer was added to each model, the parameters of which were trained and validated on 87% of images from the experimental dataset, for the task of binary classification of images as COVID-19 positive or COVID-19 negative. Each model was tested on a hold-out set consisting of the other 13% of images. Performance metrics were calculated as the average over five random 80%-20% splits of the images into training and validation sets, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Single PCX images collected from patients over 18 years of age

Exclusion Criteria:

* CT scans composed of multiple concerted X-rays
* Single PCX images collected from patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 115 COVID-19 single PCX images and 115 non COVID-19 single PCX images (230 images total), collected from 81 unique COVID-19 patients and 91 unique non COVID-19 patients.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Identification of COVID-19 | Through study completion, an average of 2 months
  Identification of COVID-19 infection from chest X-ray analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Dascena, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided